CLINICAL TRIAL: NCT02877992
Title: Development of a New Diagnostic Tool to Assess Oocyte Quality Based on Tachykinin and Kisspeptin Expression Analysis in Human Granulosa and Cumulus Cells
Brief Title: Tachykinin and Kisspeptin Expression in Human Granulosa and Cumulus Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vida Recoletas Sevilla (Other)
Responsible Party: Principal Investigator, Manuel Fernandez-Sanchez, Dr, Vida Recoletas Sevilla
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IVISEVILLA
Record Dates: First submitted 2016-08-12; First posted 2016-08-25 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Infertility
Keywords: Infertility; Tachykinin; Kisspeptin
MeSH Terms: conditions — Infertility

ARMS (5):
- Donors (Active Comparator): Oocyte donors without infertility problems
  Interventions: Procedure: Ovarian puncture
- PCOS (Experimental): Patients with Polycystic Ovary Syndrome (PCOS) according to Rotterdam criteria
  Interventions: Procedure: Ovarian puncture
- Endometriosis (Experimental): Patients with endometriosis (I-IV)
  Interventions: Procedure: Ovarian puncture
- Age (Experimental): Patients with advanced maternal age (38 years or more)
  Interventions: Procedure: Ovarian puncture
- Low ovarian response (Experimental): Patients with low ovarian response according to Bologna criteria
  Interventions: Procedure: Ovarian puncture

INTERVENTIONS:
Procedure: Ovarian puncture — Donors and patients are subjected to ovarian puncture as part of their donation procedure or IVF treatment. Oocyte are retrieved in this procedure along with granulosa and cumulus cells. Donors and patients sign an informed consent in order to donate their granulosa and cumulus cells for the study.

SUMMARY:
The purpose of this project is to study the presence of expression differences - at RNA and protein level - of different members of the tachykinin family and kisspeptin and their receptors, between fertile women and infertile patients with different etiologies.

ELIGIBILITY:
Two groups of subjects (each one with different criteria):

1. Oocyte donors

   Inclusion Criteria:
   * Age between 18 and 34 years
   * Normal caryotype
   * Normal psychological test

   Exclusion Criteria:
   * Presence of hereditary diseases
   * Beta-thalassemia
   * Cystic fibrosis
   * Human immunodeficiency virus (HIV), Hepatitis B virus (HBV), Hepatitis C virus (HCV)
2. Infertility patients

Inclusion Criteria:

* Age between 18 and 45 years
* One of the following etiologies:
* Patient with PCOS according to Rotterdam Criteria or
* Patients with endometriosis stage I-IV or
* Patients with low ovarian response according to Bologna criteria or
* Patients with advances maternal age (between 38 and 45 years)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 236 (Actual)
Dates: Start 2014-01; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Expression level of Substance P (SP) | 4 years
  Expression analysis at mRNA (mRNA = messenger ribonucleic acid) and protein level using techniques of real time quantitative PCR (PCR = polymerase chain reaction), immunocytochemistry and western blot
Expression level of neurokinin A (NKA) | 4 years
  Expression analysis at mRNA and protein level using techniques of real time quantitative PCR, immunocytochemistry and western blot
Expression level of neurokinin B (NKB) | 4 years
  Expression analysis at mRNA and protein level using techniques of real time quantitative PCR, immunocytochemistry and western blot
Expression level of hemokinin 1 (HK-1) | 4 years
  Expression analysis at mRNA and protein level using techniques of real time quantitative PCR, immunocytochemistry and western blot
Expression level of neurokinin 1 receptor (NK1R) | 4 years
  Expression analysis at mRNA and protein level using techniques of real time quantitative PCR, immunocytochemistry and western blot
Expression of neurokinin 2 receptor (NK2R) | 4 years
  Expression analysis at mRNA and protein level using techniques of real time quantitative PCR, immunocytochemistry and western blot
Expression level of neurokinin 3 receptor (NK3R) | 4 years
  Expression analysis at mRNA and protein level using techniques of real time quantitative PCR, immunocytochemistry and western blot
Expression level of kisspeptin 1 (KISS1) | 4 years
  Expression analysis at mRNA and protein level using techniques of real time quantitative PCR, immunocytochemistry and western blot
Expression level of kisspeptin 1 receptor (KISS1R) | 4 years
  Expression analysis at mRNA and protein level using techniques of real time quantitative PCR, immunocytochemistry and western blot

SECONDARY OUTCOMES:
Patient or donor age | 4 years
  Years
Patient or donor body mass index | 4 years
  kg/m2
Years of infertility | 4 years
  Number of years that the patient has been trying to have a child without success
Estradiol level (day of ovulation induction) | 4 years
  Estradiol level in blood (pg/mL), measured the day in which ovulation is induced
Progesterone level (day of ovulation induction) | 4 years
  Progesterone level in blood (ng/mL), measured the day in which ovulation is induced
Number of oocytes retrieved in the ovarian puncture | 4 years
Number of mature oocytes (metaphase II) obtained in the ovarian puncture | 4 years
Fertilization rate | 4 years
  Proportion of oocytes correctly fertilized (2 pronuclei and 2 polar bodies) after the ICSI (ICSI = intracytoplasmic sperm injection) procedure
Embryo quality | 4 years
  Embryo quality at day 3 of embryo development (of each embryo of the cohort). Quality assessed according to ASEBIR (ASEBIR = "Asociación Española para el estudio de la Biología de la Reproducción" = Spanish society for reproductive biology) criteria. Embryo quality grade A to D.
Daily and total dose of FSH (FSH = follicle stimulating hormone) | 4 years
  Daily dose of FSH for controlled ovarian stimulation. International Units (IU)
Daily and total dose of HMG (HMG = human menopausal gonadotropin) | 4 years
  Daily dose of HMG for controlled ovarian stimulation. International Units (IU)
Type of ovulation induction | 4 years
  Ovulation induction using 6500 IU of hCG (hCG = human chorionic gonadotropin) or 0.2 mg of triptorelin (Decapeptyl)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Instituto de Investigaciones Químicas, Seville
  - IVI Sevilla, Seville

REFERENCES:
- [Background] Garcia-Ortega J, Pinto FM, Fernandez-Sanchez M, Prados N, Cejudo-Roman A, Almeida TA, Hernandez M, Romero M, Tena-Sempere M, Candenas L. Expression of neurokinin B/NK3 receptor and kisspeptin/KISS1 receptor in human granulosa cells. Hum Reprod. 2014 Dec;29(12):2736-46. doi: 10.1093/humrep/deu247. Epub 2014 Oct 14. PMID 25316443
- [Result] Garcia-Ortega J, Pinto FM, Prados N, Bello AR, Almeida TA, Fernandez-Sanchez M, Candenas L. Expression of Tachykinins and Tachykinin Receptors and Interaction with Kisspeptin in Human Granulosa and Cumulus Cells. Biol Reprod. 2016 Jun;94(6):124. doi: 10.1095/biolreprod.116.139881. Epub 2016 May 4. PMID 27146034